CLINICAL TRIAL: NCT05493475
Title: Evaluation of a Novel Intervention to Prevent Polysubstance Overdoses Involving Illicit Stimulants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Nichole Michaels, Principal Investigator, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nationwide Children's Hospital
Record Dates: First submitted 2022-07-25; First posted 2022-08-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Opiate Overdose; Fentanyl Overdose; Harm Reduction
MeSH Terms: conditions — Opiate Overdose; Harm Reduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Each participant in the intervention arm will receive one-on-one education on the purpose, benefits, and limitations of fentanyl test strip (FTS) testing and undergo a brief 20-minute FTS educational intervention (including a 2-3-minute video and hands-on demonstrations on how to use FTS). They will also receive a supply of 10 FTS upon enrollment and continued supply upon request throughout the 2-year follow up period. Each participant will also receive Opioid overdose education and a naloxone kit upon enrollment and re-supply of naloxone as needed throughout the 2-year follow up period.
  Interventions: Behavioral: Fentanyl Test Strips
- Non-Intervention Arm (No Intervention): Each participant will receive Opioid overdose education and a naloxone kit upon enrollment and re-supply of naloxone as needed throughout the 2-year follow up period. Fentanyl test strip (FTS) education and a supply of FTS will be offered to participants in the non-intervention arm of the study during the final quarter of year 3.

INTERVENTIONS:
Behavioral: Fentanyl Test Strips — A brief fentanyl test strip (FTS) education intervention will be given to participants at court sites in the intervention arm after enrollment and collecting baseline data. It will be offered one-on-one with participants and will include the purpose, benefits, and limitations of FTS testing, and information on how to use FTS, interpret the results, what to do if the FTS is positive, and how to use FTS for different drug delivery methods. Participants will practice and demonstrate use of the FTS, and the short video on how to interpret the FTS will include an on-camera statement on the importance of testing for fentanyl. The video will be accessible to participants after study enrollment. Participants will be advised of the possibility of both false positive/negative results, and that the drugs may be mixed with other substances not detectable with FTS. Participants will be encouraged to practice other harm reduction strategies.
  Arms: Intervention Arm

SUMMARY:
The purpose of the study is to investigate the feasibility, acceptability, and associated benefits and harms of integrating FTS education and distribution into select courts in rural and urban communities in Ohio.

DETAILED DESCRIPTION:
Purpose: Opioid-related fatalities are a leading cause of death in Ohio and nationally, with an increasing number of overdoses attributable to fentanyl. Rapid fentanyl test strips (FTS) test for the presence of some types of fentanyl in urine samples and are increasingly being used to check illicit drugs for fentanyl before they are used. FTS use is a promising harm reduction strategy and research shows when people who use drugs (PWUD) receive a positive result, they are more likely to perform overdose risk reduction behaviors. However, access to FTS is limited, and there are barriers to the adoption of this intervention in some communities. This study will investigate FTS distribution and education as a harm reduction strategy to prevent overdoses among PWUD. Study findings will contribute valuable information about the feasibility and acceptability of integrating FTS drug checking into court sites in rural and urban communities in Ohio and help study personnel achieve the long-term goal of reducing overdose deaths.

Study Design: Court sites that volunteer to participate in the study will be randomly assigned to either the intervention or non-intervention arm of the study.

Clients in the intervention arm of the study will receive:

* One-on-one education on the purpose, benefits, and limitations of FTS testing
* A brief 20-minute fentanyl test strip educational intervention, including a 2-3-minute video and hands-on demonstrations on how to use FTS
* A supply of FTS upon enrollment and throughout the 2-year follow up period
* Opioid overdose education and a naloxone kit upon enrollment and re-supply of naloxone as needed throughout the 2-year follow up period

Clients in the non-intervention arm of the study will receive:

* Opioid overdose education and a naloxone kit upon enrollment and re-supply of naloxone as needed throughout the 2-year follow up period
* FTS education and a supply of FTS will be offered to participants in the non-intervention arm in the last year of the study

Consent: Written documentation of informed consent will be obtained from all participants.

Recruitment and Retention: Having a close partnership with the Supreme Court of Ohio will help study staff recruit and retain study participants. In addition to key informant interviews in year one and questionnaires in year three, the research team will survey court managers quarterly to collect data on the court's satisfaction with the program and identify any areas of concern. The investigators will also maintain regular communication with court personnel when the study staff are onsite.

The research team will handle all enrollment of study clients, delivery of the FTS intervention, and follow up with study participants. Court sites will be asked to provide a small space for the research team to enroll participants and provide the FTS intervention (if applicable). The sites will also be asked to refer potentially eligible individuals to the research team at times when they are on-site.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Not incarcerated at time of study enrollment
* Currently enrolled in one of the following Ohio drug courts: Criminal drug court, Veterans' court, Mental health court, Human trafficking court, Family treatment court, O.V.I. court or on probation with a participating court
* Self-reported use of illicit stimulants in the past 6 months
* Has a phone number or email address to allow for follow-up contact
* Understands English (Based on the 2012-2016 American Community Survey, only 2.4% of Ohioans 5 years and older speak English less than "very well.")

Exclusion Criteria:

- None (must meet inclusion criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Key informant interviews | Quarter 2 of Year 1
  Key informant interviews will be conducted with court personnel and peer recovery mentors who are affiliated with the court sites to discuss and obtain feedback on the intervention design and research protocols. Key informants will be asked to provide feedback on participant recruitment strategies, discuss potential barriers to the program's success, and describe any concerns with the implementation plan.
  Quantitative Data/Process Measures:
  * # interested court sites
  * # Court sites enrolled
  * # potential participants who request to enroll
  * # participants successfully enrolled
  * # people who receive FTSED and OEND at baseline
  * # replacement FTS and Naloxone kits requested/distributed
  * total # FTS and Naloxone kits distributed
  * proportion of participants in the intervention arm who complete the biweekly surveys
  * proportion of participants who complete the 6-month follow-up questionnaire
Follow-up questionnaire | Quarter 3 of Year 3
  A follow-up questionnaire will occur with intervention arm site personnel to gauge satisfaction with the program and identify any concerns.
  Quantitative Data/Process Measures:
  * # interested court sites
  * # Court sites enrolled
  * # potential participants who request to enroll
  * # participants successfully enrolled
  * # people who receive FTSED and OEND at baseline
  * # replacement FTS and Naloxone kits requested/distributed
  * total # FTS and Naloxone kits distributed
  * proportion of participants in the intervention arm who complete the biweekly surveys
  * proportion of participants who complete the 6-month follow-up questionnaire
Interview | Quarter 2 of Year 3
  Intervention arm site personnel will be interviewed to identify barriers and facilitating factors related to offering FTS education and distribution at OEND sites.
  Quantitative Data/Process Measures:
  * # interested court sites
  * # Court sites enrolled
  * # potential participants who request to enroll
  * # participants successfully enrolled
  * # people who receive FTSED and OEND at baseline
  * # replacement FTS and Naloxone kits requested/distributed
  * total # FTS and Naloxone kits distributed
  * proportion of participants in the intervention arm who complete the biweekly surveys
  * proportion of participants who complete the 6-month follow-up questionnaire
Interview | 6-month follow-up
  Intervention arm sites will be interviewed about the acceptability of the program.
  Quantitative Data/Process Measures:
  * # interested court sites
  * # Court sites enrolled
  * # potential participants who request to enroll
  * # participants successfully enrolled
  * # people who receive FTSED and OEND at baseline
  * # replacement FTS and Naloxone kits requested/distributed
  * total # FTS and Naloxone kits distributed
  * proportion of participants in the intervention arm who complete the biweekly surveys
  * proportion of participants who complete the 6-month follow-up questionnaire
Questionnaire | 6-month follow-up
  All participants (in both the intervention and non-intervention arms) will complete a questionnaire at enrollment (for the intervention group, prior to the intervention) and again at 6 months. Both questionnaires (baseline and 6 months) will include the same questions about the participant's knowledge of and self-efficacy in reducing their risk of an opioid overdose by using FTS.
Questionnaire | Quarter 3 of Year 3
  Participants in the intervention arm will be contacted biweekly for 2 years and asked if they had an overdose in the past 2 weeks and, if so, what drug they were using at the time. Intervention arm participants will be asked to notify the study team when they receive a positive FTS result. Participants in the non-intervention arm will be contacted biweekly up to a maximum of 2 years after enrollment to ask if they had an overdose in the past 2 weeks and, if so, what drug they were using at the time. Fatal overdoses among participants in the intervention and non-intervention arms of the study will be identified by reviewing death certificates issued by the Ohio Department of Health quarterly starting in Year 2.

CONTACTS AND LOCATIONS:
Overall Officials: Nichole Michaels, PhD, Principal Investigator — Nationwide Children's Hospital, Center for Injury Research & Policy; Gary Smith, MD, DRPH, Principal Investigator — Nationwide Children's Hospital, Center for Injury Research & Policy
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to de-identified IPD may be requested by qualified researchers within the scientific community after publication. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests may be submitted starting 12 months after publication and will be made available for up to 24 months.
Access Criteria: Researchers with an approved data use agreement and statistical analysis plan.